CLINICAL TRIAL: NCT02664948
Title: Early Geriatric Follow-up After Hospital Discharge in Older Acute Medical Patients - a Quasi Randomized Controlled Trial
Brief Title: Early Geriatric Follow-up in Older Acute Medical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: G-TOP-2015
Record Dates: First submitted 2015-12-17; First posted 2016-01-27 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2015-12

CONDITIONS: Geriatric Disorder
Keywords: early follow-up; geriatrics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Early geriatric follow-up after discharge from hospital in the patient's home
  Interventions: Procedure: Early geriatric follow-up after discharge
- Control group (No Intervention): Usual care with follow-up home-visits conducted by home care and the GP after discharge, if they consider it as necessary

INTERVENTIONS:
Procedure: Early geriatric follow-up after discharge — Multidisciplinary assessement and intervention by physician, nurse and physiotherapist
  Arms: Intervention group

SUMMARY:
The study is a quasi-randomized controlled trial conducted in a Danish University Hospital including older patients admitted to Emergency Department (ED). 'Early geriatric follow-up' is a multidisciplinary geriatric service provided to older patients who are discharged to their home. They receive hospital-visits by a multidisciplinary team no later than 24 hours after discharge (except on sundays). The team is consisting of a physician and a nurse both with geriatric expertise. The physician is responsible for the clinical patient care. The team is available seven days per week/12 hours per day and 24 hour on-call. In the patient's home, the team has the possibility to perform diagnosing and treatment by assessments, medication review, blood tests, subcutaneous fluid therapy, blood transfusions, intravenous antibiotics, rehabilitation and social arrangements. A discharge hand-over supports the caregivers and the GP.

DETAILED DESCRIPTION:
The study is an organizational project, which takes place in a quasi-randomized controlled design.

Every morning at the conference at the Emergency Department, patients are assessed if they are suitable for geriatric assessment and intervention and if so assigned to the Geriatric Team. Then lots are drawn by the Emergency Department's secretary (envelopes in blocks of 10) about two types of organization that is offered the patients that are admitted that day - either: 1) 'early geriatric follow-up' that comprises home visits no later than 24 hours after discharge (=intervention group), or 2) usual care after discharge with 'follow-up visits' by home care and the patient's GP, if they consider it necessary (=control group).

All the assigned patients are offered comprehensive geriatric assessment and intervention by the multidisciplinary team working in the ED consisting of a physician, nurse, and therapist, all with geriatric expertise. The assessment and intervention include evaluation of patient medication, functional ability, and social conditions.

The decision on transfer to home or to the Geriatric ward is influenced by the randomization of the day as 'early geriatric follow-up after discharge' means that more patients, with diseases that would otherwise have required treatment in hospital, can now be treated at home. Intervention patients who are considered to be too ill for treatment at home will be transferred to the Geriatric ward and then afterwards will receive 'early geriatric follow-up after discharge'.

Early follow-up starts with a visit no later than 24 hours after discharge (except for sundays). The first visit is performed by the Geriatric team and after that a tailored follow-up is performed as needed up to 30 days after discharge. The intervention can include services such as medication review, subcutaneous fluid therapy, blood transfusion, intravenous antibiotic treatment, and further examinations. The team can be contacted by phone and by e-mail. If the patient is dependent on assistance from home care, is the intervention performed in close cooperation with those. The home care is in charge of several daily observations with feedback to the team about the patient's illness and disability. In the end of the patient pathway, a discharge summary is sent to the patient's GP.

After discharge, the control group patients receive home-visits as usual by the home care and their GP, if they consider it as necessary. Before discharge, the Geriatric team has contacted the primary care and announced the discharge and sends a discharge letter. The Geriatric team is allowed to phone the patients in the control group after discharge to ensure that everything is in order and to deliver results according to hospital examinations.

ELIGIBILITY:
Inclusion Criteria:

* older patients aged 75 years or more
* admitted to Emergency Department
* one of following acute illnesses: pneumonia, delirium, dehydration, urinary tract infection, anemia, constipation, and other infection

Exclusion Criteria:

* state of terminal illness
* living outside the municipality of the hospital
* followed by other geriatric specialist teams
* included in the study within the last 30 days
* transferred to another hospital department

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2362 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Readmission (acute) | Outcome measure will be assessed as up to 30 days after discharge.(N=1330)
  Number of patients readmitted within 30 days after discharge from hospital

SECONDARY OUTCOMES:
Length of hospital stay | Outcome measure will be calculated from the date of hospital admission and up to date of discharge or date of death during hospital stay whichever came first, assessed up to 6 months (N=1330)
  Number of days from admittance at the ED to discharge from hospital
Mortality | Outcome measure will be assessed as up to 90 days after admittance to hospital (2076)
  Number of patients who died within 90 days after admittance to hospital
Patient satisfaction in a sub-group (173 patients) | Outcome measure will be assessed as up to 30 days after discharge
  14-item questionnaire based on qualitative interviews
Health costs per patient | Outcome measure will be assessed from admission as up to 30 days after discharge
  Costs used per patient at the hospital, in home care, by the GP and the pharmacy within 30 days after admittance to ED
Causes of acute readmission | Outcome measure will be assessed up to 30 days after discharge
  Assessment of avoidable and non-avoidable readmission: The causes of readmissions are assessed by three independent geriatricians through medical chart audits.
Physical functional ability | Outcome measure will be assessed 8 weeks after hospital admission(N=157)
  Assessment of Activities of Daily Living measured by Functional Recovery Score (0-100 point scale), and mobility measured by New Mobility Score (0-9 point scale)

OTHER OUTCOMES:
Avoidable readmissions | June 2014-November 2015 (N=216)
  Number of avoidable readmissions, based on a manual assessment of medical records performed by two independent reviewers

CONTACTS AND LOCATIONS:
Overall Officials: Else Marie Damsgaard, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Research Unit, Geriatric Department, Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No